CLINICAL TRIAL: NCT03144882
Title: Evaluation of Curcumin's Effect on Inflammation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TUR21324354
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Hemodialysis Complication; Hemodialysis-Induced Symptom
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): the trial group (n =35 )
  Interventions: Drug: Curcumin Pill
- placebo (Placebo Comparator): control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcumin Pill — Turmeric rhizome at first was washed and dried out in a warm and dry place for a week , then powdered rhizomes were encapsulated by Clinical Pharmacy Research Center of Shahid Beheshti University of Medical Sciences, using hard gelatin capsules. Also placebo capsules were made by the same center using Sorbitol. Curcumin level of turmeric was measured by HPTLC analysis for quantification of variability in content of curcumin
  Arms: intervention
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
Programmed ingestion of turmeric has no adverse effects and reduces plasma level of hs-CRP, IL-6 and TNF-α accompanying with increases albumin levels in hemodialysis patients. Turmeric can be considered as an effective anti-inflammatory supplement in hemodialysis patients.

DETAILED DESCRIPTION:
Hemodialysis patients over 18 years were recruited after fulfilling the inclusion criteria.Seventy-one hemodialysis patients were randomized into two groups: the trial group (n =35 ) and the controls (n =36 ); a randomization numeric table was used for allocation sequence . Trial group received turmeric and control group received placebo for 12 weeks. Biochemical determinations included levels of serum albumin (Alb), potassium (K) ,blood urea nitrogen (BUN), serum creatinine (Cr), IL-6 level, TNF- α , and liver function tests and hs-CRP at the start and end of the study were measured.

ELIGIBILITY:
Inclusion Criteria:• Males or females undergoing maintenance hemodyalisis,

* Age ≥18 year
* Clinically stable and receiving adequate hemodialysis defined by a single pool Kt/V≥1.20 or no less than 3 dialysis sessions per week with a total dialysis time ≥12 hour per week for at least 3 month before enrollment,
* Diabetic patients must be willing to commence insulin therapy if deemed necessary for plasma glucose control.

Exclusion Criteria:

* Active malignant disease (defined as less than 5 year since receiving a diagnosis of being malignancy-free)

  * Critical illness as defined by the need for respiratory or circulatory support (in an intensive care unit)
  * Active vasculitis
  * Severe congestive heart failure (New York Heart Association class IV)
  * Severe chronic systemic infectious or inflammatory disease
  * Liver disease (defined as serum alanine aminotransferase or aspartate aminotransferase levels greater than three times the upper limit of normal)
  * Known or suspected allergy to trial product(s) or related products
  * Treatment with immunosuppressive agents or receipt of any investigational drug within one month preceding screening
  * Recent or current use of anti-inflammatory corticosteroids agents
  * A scheduled renal transplantation within the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Mean Interlukin-6 Levels | one year
  blood even

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745